CLINICAL TRIAL: NCT00247910
Title: Behavioural Treatment of Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Dr. Wolfgang Linden, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C01-0175
Record Dates: First submitted 2005-10-31; First posted 2005-11-02 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2011-09

CONDITIONS: Hypertension
Keywords: hypertension, ambulatory BP, office resting BP, hydrochlorothiazide, stress reduction, self-help, psychotherapy, efficacy
MeSH Terms: conditions — Hypertension | interventions — Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Hydrochlorothiazide — Not recorded in detailed description.

SUMMARY:
The objective of the study is to determine whether psychological therapy (self-help or individualized intense stress management) is different than a single drug treatment in terms of their effectiveness for lowering blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* must be at least 19 years of age
* subjects can be male or female
* subjects must have an average resting blood pressure of >140 systolic pressure an/ or >90 diastolic pressure off anti-hypertensive medication

Exclusion Criteria:

* must not be on more than 2 blood pressure lowering drugs
* must not have known or suspected of having secondary hypertension on initial examination
* must not be pregnant or anticipating pregnancy during study period
* must not have history of allergy, hypersensitivity or intolerance to diuretics
* must not have medical condition that may result in an unacceptable risk of complications due to uncontrolled hypertension during time period of study
* must not have average resting BP readings that exceed 190 systolic, or 115 diastolic, or have two consecutive readings of 180 systolic or 110 diastolic

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2001-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Day time ambulatory BP | See description

SECONDARY OUTCOMES:
24 hour ambulatory BP, and office resting BP | See description

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Linden, PhD, Principal Investigator — University of British Columbia
Locations (1):
- UBC Hospital, Vancouver, British Columbia, Canada